CLINICAL TRIAL: NCT07348783
Title: Yogabased Movements Weekly (Online Live or Face to Face) for Primary Headaches
Brief Title: Yogabased Movements for Primary Headaches (Migraine and/or Cluster Headache) - YOURHEAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Marian Papp, Principal investigator, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNR 2025-06544-0 RCT study
Record Dates: First submitted 2025-12-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Cluster Headache - Episodic and Chronic; Migraine Headache; Migraine Headache, With or Without Aura; Migraine in Adults; Cluster Headaches and Other Trigeminal Autonomic Cephalgias; Migraine Disorder
MeSH Terms: conditions — Cluster Headache; Bronchiolitis Obliterans Syndrome; Migraine Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention yogic exercises (Experimental): Yogabased movements (online live or face to face) for primary headaches
  Interventions: Other: Intervention yoga based exercises
- No intervention - waiting list (No Intervention)

INTERVENTIONS:
Other: Intervention yoga based exercises — 8-12 weeks intervention using digital och face to face yogic exercises
  Arms: Intervention yogic exercises

SUMMARY:
Brief Summary:

Migraine and/or Cluster Headache: Study Overview

**Background:** Migraine and cluster headache are two primary headache disorders that significantly impact quality of life and functionality in those affected. According to the WHO's recurring burden of disease reports, migraine is among the neurological conditions responsible for the highest number of years lost due to illness. The headaches associated with migraine and cluster headache range from moderate to severe and cause great suffering. Available treatments do not work for everyone and are often associated with adverse side effects. Physical activity has been shown in several studies to have a positive effect on headache. Given the high prevalence of mental health issues, stress, and sleep problems within this patient group, relaxation and low-intensity exercise such as yoga-based movements (YB) could potentially help individuals improve sleep and well-being, while also providing some preventive effect on headaches.

**Hypothesis:**

Individuals with severe migraine or cluster headache have a strong need for new treatment options. Alternative therapies such as yoga-based exercises, when combined with standard medical treatment as per clinical guidelines, may positively impact:

Headache symptoms, Sleep quality and Overall life quality

* Purpose and Goals:** This randomized controlled study aims to evaluate the effect of a web-based yoga (YB) or live face to face (FTF) intervention in individuals suffering of primary headaches-mainly chronic migraine and/or cluster headache. The study will assess the effect of YB on health-related quality of life, with a focus on sleep quality and mental health as depression and anxiety. A secondary objective is to analyze changes in headache frequency, intensity, and duration associated with primary headache conditions. The RCT will also measure objective sleep and biomarkers. We are now investigating a pilot study.
* Relevance for the Patient Group:** The core objective of the project is to determine whether yoga-based exercises can serve as a complementary treatment to enhance quality of life and health in patients with severe primary headache. To ensure equal healthcare access, this intervention will be delivered in digital format and/or FTF to optimize availability and expand care for individuals with primary headache disorders. These efforts aim to improve life quality and well-being in a vulnerable patient population. Headache conditions often affect individuals in their most productive years, and many live with symptoms for decades. Both work and private life are frequently disrupted, resulting in sick leave and social isolation. Close relatives are also affected, as those suffering from headaches require more recovery time to cope with daily life. With this proposed project, we aim to use physical yoga, rooted in holistic traditional medicine, to help individuals with severe primary headache achieve better physical and mental health-particularly improved sleep quality, which in turn enhances overall life quality.

DETAILED DESCRIPTION:
Detailed Description:

Current Situation

Migraine and cluster headache are two neurological conditions characterized by recurrent attacks of severe headache. Approximately 14% of the population is estimated to suffer from migraines, while cluster headaches have a prevalence of around 0.1%. The phenotype is marked by unilateral headache attacks lasting approximately 15 minutes to three hours for cluster headache and three hours to three days for migraine. Acute treatment for migraines and cluster headaches typically involves triptans or oxygen therapy to break the attacks, and prophylactic treatment when needed.

Studies have shown that individuals with headaches experience significant impacts on quality of life and often suffer from mental health issues. Research from Karolinska Institutet and the Headache Centre in Copenhagen has demonstrated sleep disturbances among individuals with cluster headaches. Sleep-related diagnoses are also frequently reported in individuals with migraine, and migraine is more prevalent among shift workers compared to non-shift workers. Collectively, these studies indicate a strong connection between sleep problems, mental health, and headache.

The disease burden in high-frequency migraine, chronic migraine, and cluster headache is substantial, and additional alternative treatments are needed alongside standard pharmaceutical therapies. Individuals with these headache types report higher sick leave rates than the general population, and cluster headache sufferers with concurrent mental health issues show increased prevalence for long-term sick leave and disability pension.

Role of Yoga-Based Exercises (YB)

Yoga-based exercises have gained attention in healthcare and are used as complementary treatments for various conditions. Reviews and meta-analyses show effects on stress symptoms, mental states such as sleep disturbances and depression. Web-based yoga interventions have also improved sleep and stress, as well as chronic neck and back pain. Improvements have been observed in endothelial function and inflammation markers.

A review article from China indicates that physical yoga (similar to the planned intervention) appears to reduce headache intensity, duration, and frequency. Previous studies show reductions in migraine headache following yoga interventions, and smaller Indian studies report effects on headache intensity and quality of life in migraine. Research in Western contexts is limited and studies conducted in India tend to show more positive results-possibly due to higher treatment dosages or contextual influences, including placebo or Hawthorne effects.

The American Migraine Foundation recommends yoga-based exercises as a complementary treatment for stress reduction and migraine symptom management, as stress is a common migraine trigger. There is currently no research on yoga-based interventions for cluster headaches, and only a few published studies on migraines.

Traditional Medical Practices

Indian traditional medicine recommends specific exercises (e.g., inversions) for treating headaches, high blood pressure, and improving sleep quality and insomnia. Inversions appear to activate deep brain regions related to sleep and have a calming effect. Sleep disorders often trigger migraines and vice versa. Melatonin rhythms, which may be unstable in headache conditions, often stabilize following yoga-based interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed chronic migraine and/or cluster (Hortons) headache
* Men and women 18-65 years
* Diagnosed with chronic/high frequency migraine (≥15 headache days/month with at least ≥8 with migraine)
* Diagnosed with chronic cluster head ache (i.e shorter remission than 3 months per year), diagnosed according to ICHD-III criteria.
* Ability to perform yoga based moments and to give consent.
* Internet connection with computer/ipad/mobile to perform digitally/tele-health instructions
* Willing to use wristwatch for actigraphy
* Willing to leave blood samples in laboratory

Exclusion Criteria:

* Recent or planned operations during the last 6 weeks
* Drug dependence, alcohol dependence, mental disorders as psychosis, bipolar disorder, anxiety as PTSD etc)
* Parallel enrollment in other clinical trails
* Unmedicated high blood pressure, heart disease as heart failure
* Non Swedish speaking
* Not able to perform low intensity exercise at home or FTF (face to face) - both online or live.
* Participants unsure to participate due to drug addiction or other causes
* Disorientation and not able to inform regarding other serious conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Sleep quality using insomnia severity scale (ISI) | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  Primary Outcome Measure:
  Sleep quality using insomnia severity scale (ISI) [Time Frame: Baseline and 8-12 weeks after the end of the intervention, follow-up up to 24 weeks] Total score from 0-28 - a score of 0-7 no clinical insomnia, 8-14 no insomnia, 15-21 clinical insomnia moderate, 22-28 clinical insomnia severe
Quality of life - headache intensity scale (HIT-6) | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  Total score between 36-78, low scores indicates high quality of life
Dysfunctional Beliefs and attitudes about sleep (DBAS-10) | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  Measures sleep related cognitions in a VAS (visual analog)-scale. The scale identifies specific, irrationell and affective thoughts that can disturb insomnia and evaluated sleep related cognitions. Factor I (5 items) was labeled Beliefs about the Immediate Negative Consequences of Insomnia. Factor II (3 items) was labeled Beliefs about the Long-term Negative Consequences on Insomnia. Factor III was labeled Beliefs about the Need for Control Over Insomnia (2 items). Administration time 10 minutes
Actrigraph - sleep quality | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  Objective measurement of sleep using actigraphs worn on the wrist for one week at baseline and one week at the end of the study. ActTrust 2, Actiwatch or another brand is a wristwatch-like device that measures acceleration. By measuring acceleration at the wrist, an estimate of physical activity can be obtained, from which an activity pattern for a participant can be produced. This provides an objective measure of sleep duration and sleep quality. The sleep watch measures activity in general using tri-axial raw data accelerometer along with environmental light and temperature sensors and sleep is part of this through looking at reduced activity.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  Hospital Anxiety and Depression Scale (HADS) is a self-report questionnaire designed to assess anxiety and depression levels in individuals, particularly in non-psychiatric hospital settings. Structure: The questionnaire consists of 14 items, divided into two subscales: HADS-A for anxiety and HADS-D for depression. HADS uses a 4-point Likert scale (0 = not at all, 3 = most of the time), with separate scores for anxiety and depression subscales (0-21 each). Total scores range from 0 to 42, with higher scores indicating greater symptom severity. Cut-off scores for interpretation include:
  0-7: Normal. 8-10: Mild. 11-21: Moderate to severe.
Perceived stress scale (PSS-10) | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  The interpretation of perceived stress scale (PSS-10) scores is not diagnostic but provides a general sense of of perceived stress. Generally, a score between 0-13 is considered low stress, 14-26 is moderate stress, and 27-40 is high stress.
Generalized Anxiety Disorder scale (GAD-7) | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  The generalized anxiety disorder scale (GAD-7) score helps assess the severity of anxiety symptoms, with scores ranging from 0 to 21 indicating varying levels of anxiety severity.
  0 - 4: No to Minimal Symptoms - Indicates little to no anxiety symptoms. 5 - 9: Mild Symptoms - Suggests mild anxiety that may not significantly impact daily functioning.
  10 - 14: Moderate Symptoms - Indicates moderate anxiety, which may affect daily activities and quality of life.
  15 - 21: Severe Symptoms - Reflects severe anxiety that likely requires clinical intervention and support.
  Clinical Relevance A score of 10 or higher may indicate a preliminary diagnosis of Generalized Anxiety Disorder (GAD).
Nijmegen Dysfunctional breathing scale | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  The Nijmegen Questionnaire (often called the Nijmegen Dysfunctional Breathing Scale) is a validated screening tool designed to identify symptoms of dysfunctional breathing, particularly hyperventilation/overbreathing syndrome. It consists of 16 symptom items scored on a 0-4 scale, with higher scores indicating greater respiratory distress. A total score above 19-23 suggests clinically relevant breathing dysfunction. 16 items covering common symptoms such as chest pain, dizziness, blurred vision, shortness of breath, and feelings of tension.
  Each item is rated on a 5-point Likert scale: 0 = Never, 1 = Rarely, 2 = Sometimes, 3 = Often, 4 = Very often.
  19 points: Indicates possible dysfunctional breathing or hyperventilation. 23 points: Stronger indication of hyperventilation syndrome
Interleukine 6 (IL-6) | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  Biological Role IL-6 is a multifunctional cytokine produced by immune cells, endothelial cells, and glial cells. IL-6 regulates acute-phase responses, B-cell differentiation, and systemic inflammation.
  In Headache Disorders - elevated IL-6 levels have been found in migraine patients, particularly those with chronic migraine.
  IL-6 contributes to central sensitization and hypersensitivity, amplifying pain pathways.Higher circulating IL-6 before treatment has been linked to poorer outcomes in migraine preventive therapy.
  Clinical Relevance IL-6 may serve as a predictive biomarker for migraine chronification and treatment response.Its role in systemic inflammation also connects migraine with comorbidities such as obesity and cardiovascular risk.
  Healthy adults (serum/plasma) cut-off is typically <5 pg/mL above this level often indicate systemic inflammation. Migraine/Headache research show no fixed cut-off values. Studies show higher IL-6 in migraineurs compared to controls
Interleukin -1 (IL-1, especially IL-1β) | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  Interleukin-1 (IL-1, especially IL-1β) Biological Role IL-1 family cytokines (notably IL-1β) are potent mediators of inflammation. IL-1 activate endothelial cells, promote leukocyte recruitment, and stimulate nociceptors.In Headache Disorders elevated IL-1β levels have been reported in chronic tension-type headache patients.
  Salivary studies show increased IL-1β in both migraine and tension-type headache, linking it to neurogenic inflammation. IL-1β interacts with glial cells and trigeminal pathways, promoting pain transmission and headache persistence.
  Clinical Relevance IL-1β is considered a marker of neuroinflammation in headache patients. Its elevation suggests involvement in headache chronification and may help stratify patients for anti-inflammatory interventions.
  Healthy adults (serum/plasma) cut-off are usually <1-5 pg/mL, borderline elevated levels >5-10 pg/mL. IL-1 beta are often 2-3 times higher in headache migraine patients than healthy controls
Adiponectin | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  Adiponectine is an adipocyte-derived protein usually with anti-inflammatory and metabolic roles. Increased serum adiponectin levels have been observed in migraine patients compared to controls.Adiponectin can be described as paradoxical-although anti-inflammatory in metabolic contexts, it is elevated in migraine and may act as an inflammatory mediator.
  This makes it a useful biomarker for linking metabolic dysfunction (obesity, insulin resistance) with headache risk and neuroinflammation. It is anti-inflammatory in metabolic disease, but may serve as pro-inflammatory in migraine. Cut-off for men ~5-25 µg/mL (lower than women.
  Women ~7-37 µg/mL- Women have ~30-50% higher adiponectin than men, partly due to hormonal influences.
Brain-Derived Neurotrophic Factor -BDNF | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  Brain-Derived Neurotrophic Factor (BDNF) is a biomarker of neuroplasticity and pain modulation. It is a neurotrophin that supports neuronal survival and synaptic plasticity and is essential for learning and memory. BDNF is central to pain modulation and sensitization, making it a strong candidate biomarker.
  Cut-off values for healthy adults (serum/plasma)~10-50 ng/mL (varies by assay and population). ELISA assays show wide variability; levels influenced by age, sex, BMI, and physical activity.
  Low BDNF (risk marker) cut off often <10-15 ng/mL in serum/plasma Associated with depression, cognitive decline, and migraine in some studies.
  High BDNF (protective/active states) >20-25 ng/mL are linked to neuroplasticity, exercise, and better cognitive outcomes. No standardized cut-off values exist for BDNF in headache patients. Note that lower serum/plasma BDNF (<10-15 ng/mL) has been associated with migraine, depression, and poor neuroplasticity.
Melatonin (Urine, 6-sulphatoxymelatonin) | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up up to 24 weeks
  Melatonin in urine shows circadian disruption in headache patients, relevant for sleep-headache interactions.Hormone regulating circadian rhythms; urinary metabolite reflects secretion.Migraine patients show lower urinary melatonin metabolite levels compared to controls. Reduced melatonin may contribute to sleep disturbances and headache chronobiology. Supplementation has been studied as a therapeutic option. Melatonin will be measured via urinary 6-sulfatoxymelatonin. Healthy adults typically excrete 10-85 ng/mg creatinine overnight. Lower values have been reported in headache patients, reflecting circadian disruption. No standardized cut-off exists, so melatonin will be analyzed as a continuous biomarker to assess relative differences and longitudinal changes.
Headache diary - frequency of headaches | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  Headache frequency (number of days a month and number of attacks per day)
Headache diary - intensity of headaches | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  Headache intensity/pain using a visual analog scale (VAS-scale) where 0 is no pain and 100 is maximal pain.
Headache diary - duration of headaches | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  Headache duration (number of hours/minutes during an attack).
C-reactive protein (CRP) | Baseline (day 1 of the study) and 8-12 weeks after the end of the intervention, follow-up for up to 24 weeks
  C-reactive protein (CRP) will be measured in serum/plasma as a marker of systemic inflammation. Normal values are typically <3 mg/L. Levels between 3-10 mg/L indicate mild inflammation, >10 mg/L indicate clinically significant inflammation, and >100 mg/L suggest severe infection or inflammatory response. CRP will be used to assess inflammatory status and its relationship to headache and sleep outcomes.
  Inflammation marker: CRP is sensitive but non-specific; it does not identify the cause of inflammation, only its presence and intensity.
  Headache/sleep studies: Elevated CRP has been linked to poor sleep quality, migraine, and stress-related disorders

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Huddinge, Sweden